CLINICAL TRIAL: NCT06431321
Title: A Pilot Cluster Randomised Controlled Trial of a Two-session Parent Training Programme for Delivery to Caregivers of Children Enrolled in Early Childhood Development in Harare, Zimbabwe
Brief Title: Evaluation of a 2-session Parent Training Programme for Caregivers of Younger Children in Zimbabwe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Parenting for Lifelong Health (Unknown); Mikhulu Trust (Unknown); Clowns Without Borders South Africa (Unknown); Ministry of Primary and Secondary Education Zimbabwe (Unknown)
Responsible Party: Principal Investigator, Noreen Wini Dari, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WNDNOR001
Record Dates: First submitted 2024-05-08; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Child Maltreatment
Keywords: Child Maltreatment; Parenting; Violence Against Children (VAC); Prevention; Parenting Intervention; Early Childhood Development (ECD)

STUDY DESIGN:
Intervention Model Description: Each study arm will have 8 schools Schools will be randomly assigned to the study arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Research assistants and the statistician will be blinded until the analyses are completed. The randomisation process is concealed from research assistants in order to avoid experimenter bias. Complete statistical analysis plans will be prepared before the data is locked, and analysis tactics are predetermined. Until the data are finalised, the study statistician will not be aware of the treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent training intervention (Experimental): The Tabudirira Parenting Intervention for Early Childhood Development will be delivered to parents of children aged 4-5 years in Harare, Zimbabwe. Trained facilitators will deliver the programme face to face, and a group of 15 parents will have 3 facilitators. The facilitators comprise of teachers working as guidance and counselling coordinators and psychology graduates. The programme consists of 2 sessions that will be delivered once a week over 2 weeks, with each session lasting 2.5 to 3 hours. The session will have various activities which focus on learning from each other and practising positive parenting behaviours. At the end of each session, parents will receive a home activity which allows them to practise the content taught during the session. At the end of session 2 parents will receive a parent handbook with the summary of the 2 sessions. Schools will be used as venues and the facilitators will receive ongoing mentoring and coaching during programme delivery.
  Interventions: Behavioral: Tabudira Parenting Intervention for Early Childhood Development
- Control (Active Comparator): The control group (8 groups with 15 parents each) will receive a one-hour session on nutrition with facilitators trained by a nutritionist focusing on children aged 4-7 years. The parents will also receive a nutrition handbook. Zimbabwe is faced with the triple burden of malnutrition: underweight, micronutrient deficiencies and overweight. There is an ongoing need to protect and promote diets, services and practices through a multi-systems approach that supports optimal nutrition, growth, and development for all children, using a parent support group can help achieve the goal. The nutrition programme has no components of positive parenting or links to the reduction of violence against children but will serve as a placebo control for the attention received by parents.
  Interventions: Other: Nutritional guide for younger children

INTERVENTIONS:
Behavioral: Tabudira Parenting Intervention for Early Childhood Development — 2 session programme delivered weekly over 2 weeks using group-based delivery aimed at reducing child maltreatment, improving parenting behaviours and parent's mental health.
  Other Names: Parenting for Lifelong Health Young Children combined with Mikhulu Trust Book Sharing Programme - 2-Session Version
  Arms: Parent training intervention
Other: Nutritional guide for younger children — 2 session programme delivered weekly over 2 weeks aimed at providing parents with nutritional education to help provide maximum nutrition to the growing child
  Arms: Control

SUMMARY:
A pilot, exploratory cluster Randomised Controlled Trial (RCT) with two arms will be conducted to test a two-session parent training programme for caregivers of children enrolled in early childhood development classes in Harare Zimbabwe. The Parenting for Lifelong Health programme for Young Children together with the Mikhulu Trust Book Sharing Programme for Young Children will be adapted into a two-session version programme named Tabudirira Parent Training Intervention for Early Childhood Development.

The RCT aims to assess the following objectives:

Can the programme reduce child maltreatment? Does the intervention improve parent-child engagement with reading material? How best can the 2-session programme delivery be optimised?

DETAILED DESCRIPTION:
A pilot, exploratory cluster Randomised Controlled Trial (RCT) with two arms will be conducted to test a two-session parent training programme for caregivers of children enrolled in early childhood development classes in Harare, Zimbabwe. The Parenting for Lifelong Health programme for Young Children together with the Mikhulu Trust Book Sharing Programme for Young Children will be adapted into a two-session version programme named Tabudirira Parent Training Intervention for Early Childhood Development.

The RCT aims to assess the following objectives:

Can the programme reduce child maltreatment? Does the intervention improve parent-child engagement with reading material? How best can the 2-session programme delivery be optimised?

The RCt will have 2 arms with 120 caregivers /arms. The intervention will be a 2-session parent training programme while the control is a 2-session nutrition knowledge dissemination workshop delivered over 2 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above.
* Be a caregiver to a child enrolled in Early Childhood Development Grade A at a school in Harare Northern Central School district.
* Live with the child for a minimum of 5 days/ week.
* Provide informed consent before any study proceedings.

Exclusion Criteria

* Aged below 18
* A child enrolled in a school outside Harare Northern Central School District
* Child not enrolled in Early Childhood Development Grade A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06-07 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency of child maltreatment: | 6 weeks
  The International Child Abuse Screening Tool-Trial version (ICAST-T) measures the occurrence of respondents' discipline behaviour towards the child

SECONDARY OUTCOMES:
Changes in attitudes towards harsh parenting | 6 weeks
  Changes in attitudes towards harsh parenting will be measured using two items from the ICAST-T measure used in measuring the primary outcome. The questions will seek to understand parental attitudes towards harsh discipline for example: In the past 6 weeks, how often did physical discipline seem like the only option for stopping bad behaviour?
Changes in not knowing what to do when a child misbehaves | 6 weeks
  will be measured using 1 item from the ICAST-T the question: In the past 6 weeks, how often did you not know what to do when your child misbehaved
Spending time with child, praising, naming emotions | 6 weeks
  The Parenting Young Children Questionnaire (PARYC) has 9 items that contain statements of parenting behaviours that caregivers rate on a Likert scale from 1 (not at all) to 7 (most of the time). Two dimensions of the PARYC will be measured: Supporting Good Behaviour (e.g., "Notice/Praise good behaviour") and Setting Limits (e.g., "Stick to your rules"). The items included in the current questionnaire (Cronbach alpha 0.86). are informed by the metric invariance analysis of the measure done in a preceding study, pending publication. The preceding study measured the prevalence of violence against children and its correlates. The highest possible score is 63 indicating more parent-child engagement compared to the lowest possible score of 9 indicating fewer parent-child engagements.
Changes in time spent engaging the child in book sharing | 6 weeks
  Two items, similar in structure to those in the PARYC, will be used to assess this e.g. How often do you spend time book sharing with your child?
Changes in caregiver mental health | 6 weeks
  The Shona Symptoms Questionnaire (SSQ-14) will be used to assess parental mental health before and after the programme. The SSQ is a 14-item screening tool for common mental disorders and has a reliable internal consistency (0.85). It asks about symptoms such as thinking too much, failing to concentrate, work lagging, insomnia, suicidal ideation, unhappiness and so on, over 1 week. Highest total possible score of 14 indicates floundering parental mental health while a score of 0 indicates flourishing parental mental health
Changes in work-family conflict | 6 weeks
  The Multidimensional Measure of Work-Family Conflict (MMWFC) measures work-family conflict on three constructs: time, strain and behaviour. The scale has 12 items, with responses on a 7-point Likert scale ranging from strongly disagree to strongly agree. The following are examples of items in the questionnaire: my work keeps me from my family activities more than I would like, I am often stressed from my family responsibilities, and I have a hard time concentrating on my work. The internal reliability was 0.92 in phase 1. The highest possible score is 84 indicating increased work-family conflict compared to 12 which is the lowest possible score indicating better work-family balance.
Changes in Knowledge of Child nutrition | 6 weeks
  : Four questions will be adapted from the Food and Agriculture Organisation of the United Nations guidelines for assessing nutrition-related knowledge, attitudes, and practices. The questions will assess the practices of the child's intake of healthy (2 items) and unhealthy snacks (2 items): How many times a day does your child eat candy? The items will be measured on a 6-point Likert scale ranging from Never to 6 times a day. The healthy eating scores will be reverse scored. The highest possible total is 24 indicating poor snacking practices compared to the lowest possible score of 4 for healthy snacking practices.

OTHER OUTCOMES:
Implementation Outcomes | 6 weeks
  Barriers and enablers to delivery Barriers and enablers to parent engagement (attendance, homework completion)

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Wini Dari, MSc, Principal Investigator — University of Capetown
Locations (1):
- Harare Northen Central School District, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Ziva Hub Anonymised Individual Participant Data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2026
Access Criteria: Open
URL: https://zivahub.uct.ac.za/